CLINICAL TRIAL: NCT00588887
Title: Total Knee Replacement With Duracon® and Vanguard™ Prostheses
Status: Terminated | Type: Observational
Sponsor: Biomet Orthopedics, LLC (Industry)
Collaborators: New Lexington Clinic (Other)
Responsible Party: Sponsor
Organization: Zimmer Biomet (Industry)
Other Study IDs: 105-U-014
Record Dates: First submitted 2007-12-21; First posted 2008-01-09 (Estimated); Last update posted 2017-06-21 (Actual); Status verified 2017-06

CONDITIONS: Degenerative Arthritis; Osteoarthritis; Rheumatoid Arthritis; Knee Arthritis
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1
  Interventions: Device: Duracon®
- 2
  Interventions: Device: Vanguard™

INTERVENTIONS:
Device: Duracon® — This group utilizes the Duracon® prostheses for total knee replacement.
  Groups: 1
Device: Vanguard™ — This group will utilize the Vanguard™ prostheses for total knee replacement.
  Groups: 2

SUMMARY:
The purpose of this study is to compare range of motion, Knee Society Scores, and duration of surgery for different total knee prostheses.

ELIGIBILITY:
Inclusion Criteria:

* Patients with painful and disabled knee joint resulting from osteoarthritis, rheumatoid arthritis, traumatic arthritis where one or more compartments are involved.
* Patients requiring correction of varus, valgus, or posttraumatic deformity.
* Patients requiring correction or revision of unsuccessful osteotomy, arthrodesis, or failure of previous joint replacement procedure.

Exclusion Criteria:

* Patients with infection, sepsis, or osteomyelitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include patients requiring total knee replacement.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2005-06; Primary Completion 2008-02 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Range of motion, Knee Society Score, Duration of surgery | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Biomet Orthopedics, Inc., Warsaw, Indiana, United States